CLINICAL TRIAL: NCT00244595
Title: A Multicenter, Multinational, Open-Label Study of the Efficacy, Safety, and Pharmacokinetics of Candesartan Cilexetil in Hypertensive Paediatric Subjects 6 to < 17 Years of Age
Brief Title: Efficacy, Safety, & Pharmacokinetics of Candesartan Cilexetil in Hypertensive Paediatric Subjects 6 to < 17 Years of Age
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D2451C00001; 261B
Record Dates: First submitted 2005-10-25; First posted 2005-10-27 (Estimated); Last update posted 2009-12-09 (Estimated); Status verified 2009-12

CONDITIONS: Hypertension
Keywords: Pediatric hypertension; Hypertension in children
MeSH Terms: conditions — Hypertension

INTERVENTIONS:
Drug: candsartan cilexetil

SUMMARY:
The objectives of this study are to describe candesartan cilexetil antihypertensive effects in terms of achieved blood pressure and hypertension control rates and the relationship between subject characteristics and antihypertensive efficacy, and between antihypertensive therapy (candesartan cilexetil dose and add-on treatments) and efficacy over a 1 year treatment period in hypertensive children ages 6 to < 17 years; to describe growth in terms of height and weight in the study population; to describe change in neurocognition as assessed by the Full Scaled IQ score in a subset of study subjects; to determine the pharmacokinetics of candesartan in hypertensive paediatric subjects ages 6 to < 17 years; and to describe safety including adverse events and adverse events necessitating study drug discontinuation including dose level and dose duration relationships and growth over a 1 year period in hypertensive children age 6 to < 17 years.

ELIGIBILITY:
Inclusion Criteria:

* The subjects must have fulfilled the eligibility criteria for and have participated in Study 261A or did not participate in Study 261A but meet the following criteria:
* Diagnosed and untreated hypertension, or
* Diagnosed and treated, but off antihypertensive treatment for at least 2 days with a mean sitting systolic blood pressure and/or sitting diastolic blood pressure ≥ 95th percentile and ≤ 20 mm Hg (systolic) and/or 10 (diastolic) mm Hg above the 95th percentile based on height-adjusted charts for age and gender.
* Females of childbearing potential (post-menarche), must have a negative urine pregnancy test and adhere to a pregnancy prevention method (abstinence, a barrier method plus a spermicidal foam or an oral or implanted contraceptive).
* A signed informed consent by a parent or a legal guardian and an assent form signed by the subject (if applicable).

Exclusion Criteria:

* Any situation, clinical condition or laboratory abnormality that, in the opinion of the investigator or sponsor, may interfere with the subject's participation in the study or would pose a significant risk to the subject or interfere with the assessment of safety and efficacy endpoints.
* Hypertension secondary to coarctation of the aorta, pheochromocytoma, hyperthyroidism, Cushing's syndrome, or medications (eg: corticosteroids).
* Known history of bilateral renal artery stenosis, unilateral renal artery stenosis or a renal transplant.
* Glomerular filtration rate < 50 mL/min based on an estimated value using the Schwartz Formula.
* Nephrotic syndrome not in remission.
* Insulin dependent diabetes mellitus.
* Known bleeding, coagulation, or platelet disorder that could interfere with blood sampling.
* Clinically significant valvular heart disease.
* Clinical diagnosis of heart failure.
* Clinically significant arrhythmia (eg, any arrhythmia requiring medical therapy or that causes symptoms).
* Second or third degree AV block.
* Pregnant or breast-feeding an infant.
* Impaired liver function defined as either acute liver disease or chronic liver disease with persistent liver enzyme values greater than 1½ times the upper limit of the reference range for AST or ALT.
* Known hypersensitivity to ARBs.
* Unable to be off antihypertensive medication (diuretics, beta blockers, ACE Inhibitors, etc) for 6-weeks.
* Inability to discontinue medications which may contribute to elevated blood pressure e.g. systemic corticosteroids.
* Currently using, or used within 14 days prior to receiving double-blind medication, any concomitant medications which in the opinion of the investigator could negatively affect the subject.
* Unable or unwilling to comply with the study requirements including blood sampling and swallowing study drug tablets.
* Received an investigational agent within 30 days prior to receiving study medication (except in Study 261A).
* Alcohol or drug abuse.

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 235
Dates: Start 2003-09; Study Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
- Achieved sitting, trough, systolic blood pressure summarized over time and at Week 52 & the mean of the last two measures.
- The measure of effect is the mean value and the corresponding descriptive statistics.
- Additional measures include mean diastolic blood pressure, and the proportion of subjects meeting 'controlled' criteria.

SECONDARY OUTCOMES:
- Subject and baseline characteristics, antecedent treatment (eg, in 261A, an double-blind placebo-controlled efficacy study that is described elsewhere)
- The relationship to efficacy measures
- The relationship of antihypertensive treatment (candesartan cilexetil dose; add on therapy) and achieved blood pressure.

CONTACTS AND LOCATIONS:
Overall Officials: AstraZeneca Atacand Medical Science Director, MD, Study Director — AstraZeneca
Locations (44):
- United States (37):
  - Research Site, Phoenix, Arizona
  - Research Site, Beverly Hills, California
  - Research Site, Los Angeles, California
  - Research Site, Madera, California
  - Research Site, Yuba City, California
  - Research Site, Newark, Delaware
  - Research Site, Wilmington, Delaware
  - Research Site, Miami, Florida
  - Research Site, Athens, Georgia
  - Research Site, Augusta, Georgia
  - Research Site, Chicago, Illinois
  - Research Site, Park Ridge, Illinois
  - Research Site, Louisville, Kentucky
  - Research Site, Ann Arbor, Michigan
  - Research Site, Jackson, Mississippi
  - Research Site, Port Gibson, Mississippi
  - Research Site, St Louis, Missouri
  - Research Site, Las Vegas, Nevada
  - Research Site, Paterson, New Jersey
  - Research Site, Brooklyn, New York
  - Research Site, New Hyde Park, New York
  - Research Site, The Bronx, New York
  - Research Site, Charlotte, North Carolina
  - Research Site, Winston-Salem, North Carolina
  - Research Site, Cincinnati, Ohio
  - Research Site, Cleveland, Ohio
  - Research Site, Columbus, Ohio
  - Research Site, Portland, Oregon
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Pittsburgh, Pennsylvania
  - Research Site, Charleston, South Carolina
  - Research Site, Beaumont, Texas
  - Research Site, Houston, Texas
  - Research Site, Salt Lake City, Utah
  - Research Site, Charlottesville, Virginia
  - Research Site, Norfolk, Virginia
  - Research Site, Charleston, West Virginia
- Research Site, Ghent, Belgium
- Hungary (3):
  - Research Site, Budapest
  - Research Site, Miskolc
  - Research Site, Szeged
- Slovakia (3):
  - Research Site, Bratislava
  - Research Site, Martin
  - Research Site, Trnava